CLINICAL TRIAL: NCT02416999
Title: Ultra-low Dose Bevacizumab Plus Temozolomide for Recurrent High-grade Gliomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Yanda Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YDCR-2015-001
Record Dates: First submitted 2015-04-01; First posted 2015-04-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent High-grade Glioma
Keywords: glioma; high-grade glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patient group (Experimental)
  Interventions: Drug: Ultra-low dose Bevacizumab; Drug: Temozolomide

INTERVENTIONS:
Drug: Ultra-low dose Bevacizumab
  Other Names: BVZ
Drug: Temozolomide
  Other Names: TMZ

SUMMARY:
This study is to evaluate the effectiveness of ultra-low dose Bevacizumab plus Temozolomide for recurrent high-grade gliomas.

DETAILED DESCRIPTION:
This trial is aimed at evaluating the effectiveness of ultra-low dose Bevacizumab plus Temozolomide for recurrent high-grade gliomas. And, this trial is approved by medical ethics committee of Hebei Yanda Hospital.Researchers will conduct thsi trial from 2015/05 to 2018/05, and 30 recurrent high-grade glioma patients will be recruited. Patients who are recruited will get treatment of ultra-low dose Bevacizumab plus Temozolomide in ether Hebei Yanda Hospital or Beijing Tiantan hospital, and get follow-ups from clinicians.

ELIGIBILITY:
Inclusion Criteria:

* High grade glioma was diagnosed by post-operation pathological method, and shows a relapse.
* Before included, the patient needs imageological examinations, and the diameter of contrast enhancing area is bigger than 1cm, PET or MRS results show positive features.
* The age of patient should be between 18 years old and 70 years old.
* The condition of the patient permits the treatment of ultra-low dose Bevacizumab plus Temozolomide.
* The patient is informed consent,and willing to join in this research.

Exclusion Criteria:

* The diagnosis is not recurrent high-grade glioma.
* The diagnosis of high-grade glioma was not established by pathological method.
* The results of imageological examinations do not meet the standard of including.
* The age of the patient does not meet the requirement of this research.
* The condition of the patient does not permit the treatment of ultra-low dose Bevacizumab plus Temozolomide.
* There are other conditions that the clinicians believe that the treatment of ultra-low dose Bevacizumab plus Temozolomide is not appropriate for the patient.
* The patient is not willing to join in this research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
6-month survival rate of recurrent glioblastoma multiforme patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 6 months
12-month survival rate of recurrent WHO-III glioma patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 12 months

SECONDARY OUTCOMES:
Overall survival of recurrent glioblastoma multiforme patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 6 months or later, up to 12 months
Overall survival of recurrent WHO-III glioma patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 12 months or later, up to 24 months
Progression free survival of recurrent glioblastoma multiforme patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 6 months or later, up to 12 months
Progression free survival of recurrent WHO-III glioma patients under ultra-low dose Bevacizumab plus Temozolomide treatment | 12 months or later, up to 24 months
6-month life quality as measured by European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30 and EORTC QLQ-BN20 together) | 6 months
12-month life quality as measured by European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30 and EORTC QLQ-BN20 together) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jisheng Wang, MD, Principal Investigator — Beijing Tiantan Hospital; Nan Ji, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Hebei Yanda Hospital, Sanhe, Hebei